CLINICAL TRIAL: NCT05275543
Title: Robot Rehab: Animal Assisted Interactions With a Robotic Baby Harp Seal During Inpatient Pediatric Rehabilitation
Brief Title: Robot Rehab: AAI With Robot During Inpatient Pediatric Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0010-22-EP
Record Dates: First submitted 2022-02-25; First posted 2022-03-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-03

CONDITIONS: Pediatric ALL; Child, Hospitalized; Physical Therapy Modalities; Occupational Therapy; Animal Assisted Therapy
Keywords: Robot; Animal Assisted Interaction; Hosptilization; Rehabiliation; Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with Repeated Measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Physical and Occupational Therapy with Paro Robot (Experimental): 10-30 minute semi-structured, prescriptive therapy sessions with Paro robot focused on the categories of 1) speech; 2) balance and endurance; 3) memory; 4) self-esteem; 5) fine motor; 6) sensory stimulation
  Interventions: Device: Paro Robot
- Physical and Occupational Therapy without Paro Robot (No Intervention): 10-30 minute semi-structured, prescriptive therapy sessions without Paro robot focused on the categories of 1) speech; 2) balance and endurance; 3) memory; 4) self-esteem; 5) fine motor; 6) sensory stimulation
- Parents/Guardians of Hospitalized Children who use Paro Robot (Experimental): Parents/guardians of hospitalized children who are assigned to the following arm "Physical and Occupational Therapy with Paro Robot"
  Interventions: Device: Paro Robot
- Parents/Guardians of Hospitalized Children who do not use Paro Robot (No Intervention): Parents/guardians of hospitalized children who are assigned to the following arm "Physical and Occupational Therapy with out Paro Robot"

INTERVENTIONS:
Device: Paro Robot — Device: PARO therapy seal PARO, a baby harp seal, is an advanced interactive, therapeutic medical robot developed by AIST, a leading Japanese industrial automation pioneer. It allows the documented benefits of animal therapy to be administered to patients in environments such as hospitals and extended care facilities where live animals present treatment or logistical difficulties.
  Arms: Parents/Guardians of Hospitalized Children who use Paro Robot; Physical and Occupational Therapy with Paro Robot

SUMMARY:
The purpose of this study is to:

Aim 1: Evaluate the feasibility [consent and refusal rates, attrition rates, length, and number of completed therapy sessions], and acceptability [interviews with children and guardians, overall patient and guardian satisfaction] during inpatient physical therapy (PT) and occupational therapy (OT) sessions. Hypothesis: Animal-assisted interaction (AAI) with Paro, a robotic baby harp seal, during pediatric inpatient PT/OT sessions will be feasible and acceptable.

Aim 2: Assess preliminary efficacy of AAI during PT/OT sessions with Paro on behavior (anxiety and affect) and motivation to participate in rehabilitation in hospitalized children. Hypothesis: Children who use Paro will demonstrate less anxiety, more positive affect, and greater motivation to participate in therapy than those who do not use Paro.

Aim 3: Test the stress, anxiety, and depression levels of parents/guardians of children who use Paro inpatient physical and occupational therapy sessions. Hypothesis: In addition, parents and guardians of children that use Paro will report less stress, anxiety, and depression compared to parents/guardians of children that do not use Paro.

DETAILED DESCRIPTION:
Animal Assisted Interactions (AAIs) are interventions that intentionally incorporate animals as part of a therapeutic process to promote human health, learning, and well-being. In general, domestic and farm animals such as dogs, cats, birds, equines, guinea pigs, rabbits, llamas, sheep, goats, and pigs are predominantly featured in AAI programs. Animals can be observed, held, and petted, or more actively integrated into specific therapy activities such as brushing with different tools to encourage range of motion and fine motor coordination. AAIs also promote exercise through tandem walking with the animals. Recent literature indicates that AAI can improve reality orientation and attention span, eliminate the sense of isolation, reduce stress and anxiety, enhance communication, promote positive social interactions, and enhance overall quality of life. The use of AAI in hospitalized children has the potential to engage patients, family members, and healthcare staff in an innovative, holistic approach to recovery.

While additional research is warranted to further explore the potential impact of AAI on a variety of clinically meaningful patient outcomes, the highly technical, fast-paced hospital environment and the immunocompromised health statuses of many acutely ill hospitalized patients greatly limit the exploration of AAI in inpatient settings. A new frontier in animal robotics opens a vast array of opportunities to implement AAI in hospitalized populations. Robot animals may be just as effective as live animals and may provide even more flexibility and tailoring to meet the needs of diverse situations that arise in the hospital. In addition, the infection control risk that live animals pose to hospitalized patients may be significantly lessened.

For this study, the investigators plan to conduct a two-armed randomized controlled trial with repeated measures. Hospitalized pediatric patients will participate in semi-structured, prescriptive physical and occupational therapy sessions on the categories of: 1) speech; 2) balance and endurance; 3) memory; 4) self-esteem; 5) fine motor; 6) sensory stimulation. Intervention group subjects (n=30) will participate in 10-30 minute therapy sessions with Paro, a therapeutic robotic baby harp seal. Control group subjects (n=30) will participate in 10-30 minute therapy sessions without Paro.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18
* admitted to any of the five inpatient units at Children's Hospital and Medical Center, Omaha, NE
* have an available parent or guardian
* have an active consult request for PT or OT
* awake, alert, able to follow commands
* not delirious
* able to understand English
* free from significant vision or hearing deficits
* able to verbalize.

Exclusion Criteria:

* Have a pacemaker
* have airborne, enteric, or enhanced contact precautions
* wounds without a covering dressing or a dressing that is visibly soiled
* known adverse psychological reactions to animals
* excessive secretions via nose or mouth
* report feeling nauseated
* shows signs of acute agitation (yelling, screaming, moaning, or is otherwise inconsolable).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Pain: Wrong-Baker FACES pain rating scale | Change from before therapy session to immediately after therapy session is completed
  The scale shows a series of faces ranging from a happy face at 0 which represents "no hurt" to a crying face at 10 which represents "hurts worst." Based on the faces and descriptions, the patient chooses the face that best describes their level of pain.
Anxiety: Children's Anxiety Meter-State (CAM-S) | Change from before therapy session to immediately after therapy session is completed.
  The CAM scale is drawn to resemble a thermometer with a bulb at the bottom and horizontal lines at intervals going up to the top. The child is instructed to indicate with a line how the child feels from from the bottom of the thermometer (not worried or nervous) to the top (very worried or nervous).
Intervention Acceptability | Within 1 week of study completion
  Patient Satisfaction Measure: Investigator-developed Satisfaction Measure contains one item which asks the participants to rank their satisfaction with the intervention from 1-5 (not at all - very much)
Hospital Acquired Infections-Central Line Associated Blood Stream Infections (CLABSI) | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Rates of Central Line Associated Blood Stream Infections (CLABSI) will be collected from the electronic medical record.
Hospital Acquired Infections-Catheter-Associated Urinary Tract Infections (CAUTI) | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Rates of Catheter-Associated Urinary Tract Infections (CAUTI) will be collected from the electronic medical record.
Hospital Acquired Infections-Enteroviruses | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Rates of Enteroviruses will be collected from the electronic medical record.
Hospital Acquired Infections-Influenza | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Rates Influenza will be collected from the electronic medical record.
Hospital Acquired Infections-Multi-Drug Resistant Organisms | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Rates of Multi-Drug Resistant Organisms will be collected from the electronic medical record.
Hospital Acquired Infections-Surgical-Site Infections (SSI) | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Surgical-Site Infections (SSI) will be collected from the electronic medical record.
Hospital Acquired InfectionsVentilator-Associated Pneumonia (VAP) | Chart review will be conducted from the first day the patient is enrolled until 1 week after study completion.
  Rates of Ventilator-Associated Pneumonia (VAP) will be collected from the electronic medical record.
Sedation Exposure | 4 hours after each individual session
  Sedative and analgesic medications will be abstracted from the electronic medical record (EMR) in order to calculate sedation frequency for 4 hours after each PT/OT session in which PARO was used.
Microbial Contamination Screening | Completed immediately after each individual session
  The ATP Monitoring with SystemSURE Plus Process uses a process which monitors levels of ATP Bioluminescence The investigators will implement established cleaning protocols and then measure ATP before the PT/OT session by swabbing PARO on the following areas: head, right flipper, left flipper, bottom [by on/off switch], top left back area, top right back area, stomach [underneath].
Activity performance form | Immediately after each intervention therapy sesison
  The Activity Performance Form is an investigator developed measure that assesses the length of each therapy session (in minutes), the time to the patient's first out of bed movement, as well as the number and types of range of motion exercises performed (Passive, Active assist, and Active)
Physiologic variables-Blood Pressure | Change from before therapy session to immediately after therapy session is completed
  Blood Pressure (systolic & diastolic)
Physiologic variables-Respiratory Rate | Change from before therapy session to immediately after therapy session is completed
  Respiratory Rate
Physiologic variables | Change from before therapy session to immediately after therapy session is completed
  Oxygen Saturation
Opinion on Pets | Prior to the start of the first therapy session.
  18-item instrument with seven-point Likert scale (1-strongly disagree to 7-strongly agreed) designed to measure the favorableness of attitudes toward pets. Minimum Score = 18; Maximum score = 126. The higher the score, the more favorable a patient feels towards pets.
Parent/Guardian Stress | Change from the start of the first therapy session to the end of the final therapy session.
  42-item instrument with a five-point Likert scale designed to measure stress in parents whose child has a chronic illness or requires prolonged medical monitoring. It includes four domains or subscales. Minimum Score = 42; Maximum Score = 210. Higher scores indicate higher stress.
Parent/Guardian Anxiety and Depression | Change from the start of the first therapy session to the end of the final therapy session.
  Parent/Guardian anxiety and depressive symptoms as measured by the Hospital Anxiety and Depression Scale (HADS). Two sub-scales (Anxiety & Depression) scored separately. Minimum Score = 0; Maximum Score = 21. Higher score = higher anxiety and/or depression
Mood/Affect | Change from the start of the first therapy session to the end of the final therapy session.
  The PANAS-10 is a 10-item instrument that asks the child to rate adjectives of varying mood states according to how often the child feels joyful, cheerful, happy, lively, proud, miserable, mad, afraid, scared, and sad. The item response uses a five-point Likert scale ranging from 1 ("very slightly or none at all") to 5 ("extremely"). Minimum score = 10; Maximum score = 50. The higher the score, the better a child's mood/affect
Motivation to Participate in Therapy | Immediately after each therapy session.
  19-item scale with a six-point smiley-face scale and two open-ended questions to measure motivation from a child's perspective. It has six subscales (interest/enjoyment, competence, relatedness, autonomy, value/usefulness, and effort/importance).tems in each subscale are totaled and divided by the number of items to obtain an average score per subscale. The total scores in each subscale are added to obtain and overall motivation score. Higher scores within each subscale indicate a higher level of the concept in the subscale, whereas lower scores indicate the opposite. Thus, the scores indicate differences in the quality and type of motivation for the child. In addition, a higher total score indicates greater levels of motivation, overall.

CONTACTS AND LOCATIONS:
Overall Officials: Breanna D Hetland, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Children's Hosptial and Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fine AH. Handbook on Animal-Assisted Therapy: Theoretical Foundations and Guidelines for Practice. 4th ed. Burlington, MA: Academic Press; 2015
- [Background] Bailey T, Christenson G, Lust K. The role of an animal-assisted interaction (AAI) program as a means of reducing stress and anxiety within a college community. Oxford, UK: Inter-Disciplinary Press.
- [Background] Bailey T. Animal-assisted interactions (AAI): a creative modality to support youth with depression. In: Brooke SL, Myers CE, eds. The Use of the Creative Therapies in Treating Depression. Springfield, IL: Charles C. Thomas; 2015:269.
- [Background] Burres S, Edwards NE, Beck AM, Richards E. Incorporating Pets into Acute Inpatient Rehabilitation: A Case Study. Rehabil Nurs. 2016 Nov;41(6):336-341. doi: 10.1002/rnj.260. Epub 2016 Mar 9. PMID 26956570
- [Background] Hetland B, Bailey T, Prince-Paul M. Animal Assisted Interactions to Alleviate Psychological Symptoms in Patients on Mechanical Ventilation. J Hosp Palliat Nurs. 2017 Dec;19(6):516-523. PMID 29276432
- [Background] Templer D.I., Arikawa H. (2011) The Pet Attitude Scale. In: Blazina C., Boyraz G., Shen-Miller D. (eds) The Psychology of the Human-Animal Bond. Springer, New York, NY. https://doi.org/10.1007/978-14419-9761-6_20
- [Background] Streisand R, Braniecki S, Tercyak KP, Kazak AE. Childhood illness-related parenting stress: the pediatric inventory for parents. J Pediatr Psychol. 2001 Apr-May;26(3):155-62. doi: 10.1093/jpepsy/26.3.155. PMID 11259517
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Background] Ersig AL, Kleiber C, McCarthy AM, Hanrahan K. Validation of a clinically useful measure of children's state anxiety before medical procedures. J Spec Pediatr Nurs. 2013 Oct;18(4):311-9. doi: 10.1111/jspn.12042. Epub 2013 Jun 25. PMID 24094126
- [Background] Ebesutani C, Regan J, Smith A, Reise S, Higa-McMillan C, Chorpita BF. The 10-item positive and negative affect schedule for children, child and parent shortened versions: Application of item response theory for more efficient assessment. J of Psychopathol. Behav. Assess. 2012; 34(2), 191-203.
- [Background] Tatla SK, Jarus T, Virji-Babul N, Holsti L. The development of the Pediatric Motivation Scale for rehabilitation. Can J Occup Ther. 2015 Apr;82(2):93-105. doi: 10.1177/0008417414556884. PMID 26281433
- [Background] Tracy MF, Chlan L, Savik K, Skaar DJ, Weinert C. A Novel Research Method for Determining Sedative Exposure in Critically Ill Patients. Nurs Res. 2019 Jan/Feb;68(1):73-79. doi: 10.1097/NNR.0000000000000322. PMID 30540694